CLINICAL TRIAL: NCT03809624
Title: An Open-Label, Multicenter, First-in-Human, Dose-Escalation, Phase 1 / 2 Study of INBRX-105 and INBRX-105 in Combination With Pembrolizumab in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of INBRX-105 and INBRX-105 With Pembrolizumab in Patients With Solid Tumors Including Head and Neck Cancer
Acronym: PDL1x41BB
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Program terminated due to lack of meaningful efficacy signal.
Sponsor: Inhibrx Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Ph 1 Ph 2 INBRX-105
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Solid Tumors; Non-small Cell Lung Cancer; Melanoma; Head and Neck Squamous Cell Carcinoma; Gastric Adenocarcinoma; Renal Cell Carcinoma; Esophageal Adenocarcinoma; Nasopharyngeal Carcinoma; Oropharyngeal Carcinoma
Keywords: Solid Tumors; Lung Cancer; Melanoma; Head and Neck Cancer; Stomach Cancer; Gastric Cancer; Kidney Cancer; Renal cell carcinoma; Renal Cancer; Urothelial Carcinoma; PDL1; 41BB; PD-L1; 4-1BB; Pembrolizumab; Keytruda; Nasopharyngeal carcinoma; Oropharyngeal carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Adenocarcinoma Of Esophagus; Nasopharyngeal Carcinoma; Oropharyngeal Neoplasms; Lung Neoplasms; Head and Neck Neoplasms; Stomach Neoplasms; Kidney Neoplasms; Carcinoma, Transitional Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Single Agent Escalation (Experimental): INBRX-105 will be escalated in patients with locally advanced or metastatic solid tumors.
  Interventions: Drug: INBRX-105 - PDL1x41BB antibody
- Expansion Cohort Non-small Cell Lung Cancer (Experimental): Patients will be treated with single-agent INBRX-105 at either the MTD or RP2D.
  Interventions: Drug: INBRX-105 - PDL1x41BB antibody
- Expansion Cohort Melanoma (Experimental): Patients will be treated with single-agent INBRX-105 at either the MTD or RP2D.
  Interventions: Drug: INBRX-105 - PDL1x41BB antibody
- Expansion Cohort PD-L1 Positive Basket (Experimental): Patients with gastric or gastro-esophageal junction adenocarcinoma, renal cell carcinoma, and urothelial (transitional) cell carcinoma will be treated with single-agent INBRX-105 at either the MTD or RP2D.
  Interventions: Drug: INBRX-105 - PDL1x41BB antibody
- Expansion Cohort Nasopharyngeal or Oropharyngeal Carcinoma (Experimental): Patients with head and neck squamous cell carcinoma (NPC or OPC) will be treated with single-agent INBRX-105 at either the MTD or RP2D.
  Interventions: Drug: INBRX-105 - PDL1x41BB antibody
- INBRX-105 Escalation in Combination with Pembrolizumab (Experimental): INBRX-105 will be escalated in combination with Pembrolizumab in pateitns with locally advanced or metastatic solid tumors.
  Interventions: Drug: INBRX-105 - PDL1x41BB antibody; Drug: Pembrolizumab
- Combination Expansion Cohort Non-small Cell Lung Cancer (Experimental): CPI relapsed/refractory patients will be treated with INBRX-105 in combination with Pembrolizumab.
  Interventions: Drug: INBRX-105 - PDL1x41BB antibody; Drug: Pembrolizumab
- Combination Expansion Cohort Melanoma (Experimental): CPI relapsed/refractory patients will be treated with INBRX-105 in combination with Pembrolizumab.
  Interventions: Drug: INBRX-105 - PDL1x41BB antibody; Drug: Pembrolizumab
- Combination Expansion Cohort Cohort PD-L1 Positive Basket (Experimental): CPI-relapsed/refractory patients with head and neck squamous cell carcinoma, gastro-esophageal junction adenocarcinoma, renal cell carcinoma, and urothelial (transitional) cell carcinoma will be treated with INBRX-105 in combination with Pembrolizumab.
  Interventions: Drug: INBRX-105 - PDL1x41BB antibody; Drug: Pembrolizumab
- Combination Expansion Cohort CPI Naive Non-small Cell Lung Cancer (Experimental): CPI naive patients (PD-L1 IHC between 1 and 49%) will be treated with INBRX-105 in combination with Pembrolizumab.
  Interventions: Drug: INBRX-105 - PDL1x41BB antibody; Drug: Pembrolizumab
- Combination Expansion Cohort CPI Naive HNSCC (Experimental): CPI naive patients (PD-L1 IHC >50%) will be treated with INBRX-105 in combination with Pembrolizumab.
  Interventions: Drug: INBRX-105 - PDL1x41BB antibody

INTERVENTIONS:
Drug: INBRX-105 - PDL1x41BB antibody — The active ingredient of INBRX-105 is a recombinant, humanized, bispecific IgG antibody that targets the human programmed death-ligand 1 (PD-L1) receptor and the human 4-1BB receptor.
Drug: Pembrolizumab — Pembrolizumab 200 mg by intravenous (IV) infusion, given on Day 1 of each 21-day cycle.
  Other Names: Keytruda
  Arms: Combination Expansion Cohort CPI Naive Non-small Cell Lung Cancer; Combination Expansion Cohort Cohort PD-L1 Positive Basket; Combination Expansion Cohort Melanoma; Combination Expansion Cohort Non-small Cell Lung Cancer; INBRX-105 Escalation in Combination with Pembrolizumab

SUMMARY:
This is a first-in-human, open-label, nonrandomized, four-part trial to determine the safety profile and identify the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of INBRX-105 and INBRX-105 in combination with Pembrolizumab. INBRX-105, a next generation bispecific antibody, targets the human programmed death-ligand 1 (PD-L1) receptor and the human 4-1BB receptor. INBRX-105 provides localized conditional T-cell co-stimulation through 4-1BB agonism.

ELIGIBILITY:
Inclusion Criteria:

* Parts 1 and 3 (escalation cohorts; completed): Patients with locally advanced or metastatic non-resectable solid tumors, whose disease has progressed despite standard therapy and for whom no further standard therapy exists.
* Part 2 (expansion cohorts): Patients with non-small cell lung cancer, cutaneous melanoma, head and neck squamous cell carcinoma or solid tumors amenable to paired biopsies, with locally advanced or metastatic, non-resectable disease, which has progressed despite standard therapy or for whom no standard or clinically acceptable therapy exists.
* Part 4 relapsed or refractory to CPI cohorts: NSCLC, cutaneous melanoma, HNSCC, MSI/TMB-high or MMRd solid tumors
* Part 4 CPI naive cohorts: locally advanced or metastatic, non-resectable NSCLC or HNSCC
* Refractory or relapsed to anti-PD-1 or anti-PD-L1, and anti-CTLA4 if applicable (NOTE: For all tumor types with checkpoint inhibitor approvals) with exception of the treatment naive NSCLC cohort.
* PD-L1 positivity by immunohistochemistry (IHC): Parts 1 and 3 (escalation cohorts) PD-L1 positivity is not required. Parts 2 and 4 (expansion cohorts): Combined Positive Score (CPS) or Tumor Proportion Score (TPS) above certain thresholds as defined per protocol.
* Adequate hematologic, coagulation, hepatic and renal function as defined per protocol.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.

Exclusion Criteria:

* Prior exposure to 4-1BB agonists.
* Receipt of any investigational product or any approved anticancer drug(s) or biological product(s) within 4 weeks prior to the first dose of study drug. Exceptions: Hormone replacement therapy, testosterone, or oral contraceptives. NOTE: Previous exposure to anti-PD-L1 checkpoint inhibitor requires a minimum washout period of 24 weeks prior to the first dose of study drug.
* Hematologic malignancies (e.g., ALL, AML, MDS, CLL, CML, NHL, Hodgkin lymphoma and multiple myeloma).
* Prior or concurrent malignancies. Exception: Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessments of INBRX-105.
* Known or active primary central nervous system (CNS) tumors, leptomeningeal disease and CNS metastases. Exception: Subjects with previously treated, asymptomatic, and clinically stable CNS metastases may be allowed study entry if certain criteria apply.
* Grade ≥ 3 immune-related adverse events (irAEs) or irAE that lead to discontinuation of prior immunotherapy. Some exceptions as defined per protocol apply.
* Active autoimmune disease or documented history of autoimmune disease that required systemic steroids or other immunosuppressive medications. Certain exceptions as defined in protocol apply.
* Treatment with systemic immunosuppressive medications within 4 weeks prior to the first dose of study drug. Certain exceptions as defined in protocol apply.
* History of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV). Exceptions as defined in protocol for expansion cohorts will apply.
* History of hepatitis or cirrhosis (e.g., non-alcohol steatohepatitis, alcohol or drug-related, autoimmune, hepatitis B, or hepatitis C). Exceptions as defined in protocol for expansion cohorts will apply.
* Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment with steroids or other immunosuppressive medications.
* Clinically significant cardiac condition, including myocardial infarction, uncontrolled angina, cerebrovascular accident, or other acute uncontrolled heart disease < 3 months; left ventricular ejection fraction (LVEF) < 50%; New York Heart Association (NYHA) Class III or IV congestive heart failure; or uncontrolled hypertension.
* Active, hemodynamically significant pulmonary embolism within 3 months prior to enrollment on this trial.
* Major surgery within 4 weeks prior to enrollment on this trial.
* Anti-infectious drug treatments (i.e., antibiotics) within 4 weeks prior to the first dose of study drug.
* Prior organ allograft transplantations or allogeneic peripheral blood stem cell (PBSC) or bone marrow (BM) transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events of INBRX-105 | Up to 2-3 years
  Adverse events will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Severity of adverse events of INBRX-105 | Up to 2-3 years
  Severity of adverse events will be assessed and assigned by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of INBRX-105 | Up to 2-3 years
  The MTD and/or RP2D of INBRX-105 will be determined.

SECONDARY OUTCOMES:
Area under the serum concentration time curve (AUC) of INBRX-105 | Up to 2-3 years
  Area under the serum concentration time curve (AUC) of INBRX-105 will be determined.
Maximum observed serum concentration (Cmax) of INBRX-105 | Up to 2-3 years
  Maximum observed serum concentration (Cmax) of INBRX-105 will be determined.
Trough observed serum concentration (Ctrough) of INBRX-105 | Up to 2-3 years
  Trough observed serum concentration (Cmax) of INBRX-105 will be determined.
Time to Cmax (Tmax) of INBRX-105 | Up to 2-3 years
  Time to Cmax (Tmax) of INBRX-105 will be determined.
Immunogenicity of INBRX-105 | Up to 2-3 years
  Frequency of anti-drug antibodies (ADA) against INBRX-105 will be determined.

OTHER OUTCOMES:
Anti-tumor activity of INBRX-105 | Up to 2-3 years
  Tumor response will be determined by immune Response Evaluation Criteria in Solid Tumors (iRECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead, Study Director — Inhibrx Biosciences, Inc
Locations (23):
- United States (23):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - City of Hope at Irvine Lennar, Duarte, California
  - City of Hope, Duarte, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado Denver, Denver, Colorado
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Norton Cancer Center, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - Nebraska Cancer Specialists - Grand Island, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Providence Cancer Institute, Portland, Oregon
  - Abramson Cancer Center - University of Pennsylvania, Philadelphia, Pennsylvania
  - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - New Experimental Therapeutics of San Antonio - NEXT Oncology, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Northwest Medical Specialties, PLLC, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No